CLINICAL TRIAL: NCT07020429
Title: Efficacy and Safety of the Traditional Chinese Herbal Formula Huanjingjian Decoction in Women With Premature Ovarian Insufficiency: a Randomised Controlled Trial
Brief Title: Efficacy and Safety of Huanjingjian Decoction in Women With Premature Ovarian Insufficiency
Acronym: EAST-HOPE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Collaborators: Shanghai University of Traditional Chinese Medicine (Other); Shanghai Geriatric Institute of Chinese Medicine (Unknown); Shanghai Institute of Acupuncture and Anesthesia, Shanghai (Unknown); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Jingan Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Principal Investigator, Wei Wu, Attending Physician, Department of Anesthesiology, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202240223
Record Dates: First submitted 2025-05-16; First posted 2025-06-13 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Premature Ovarian Insufficiency
Keywords: premature ovarian insufficiency; menopause; traditional Chinese herbal formula; Huanjingjian decoction
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Hormone Replacement Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, care providers, investigators, and outcome assessors will remain blinded to the treatment allocation throughout the trial. Randomisation codes will be generated by an independent statistician who is not involved in participant recruitment. Study medications (Huanjingjian decoction and placebo) will be manufactured and packaged to be identical in appearance, taste, and packaging. Sealed envelopes containing the randomisation codes will be kept securely by the clinical trial unit and may only be opened in case of a medical emergency or a serious adverse event requiring unblinding. Furthermore, the statisticians conducting the data analysis will maintain blinding during the analysis phase, with datasets identified solely as Group A and Group B to ensure unbiased evaluation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Huanjingjian decoction + Hormone replacement therapy (Experimental): Participants in this group will receive treatment with Huanjingjian decoction in combination with hormone replacement therapy (HRT).
  Interventions: Drug: Huanjingjian decoction; Drug: Hormone replacement therapy
- Placebo + Hormone replacement therapy (Active Comparator): Participants in this group will receive treatment with hormone replacement therapy (HRT) in combination with placebo.
  Interventions: Drug: Hormone replacement therapy; Drug: Placebo

INTERVENTIONS:
Drug: Huanjingjian decoction — Participants will receive the traditional Chinese herbal formulation Huanjingjian decoction, administered at a dose of one vial (10 ml) twice daily, taken 30 minutes after breakfast and dinner. The intervention will commence immediately following the cessation of menstruation and will continue until the onset of the subsequent menstrual period. Upon the completion of each menstrual cycle, the treatment will be resumed. Each treatment course spans 28 days, with a total of three consecutive cycles administered.
  Arms: Huanjingjian decoction + Hormone replacement therapy
Drug: Hormone replacement therapy — Participants will begin oral administration of Utrogestan (estradiol valerate) on the 5th day of menstruation at a dose of 1 mg daily for 21 consecutive days. Starting from day 17 of treatment, medroxyprogesterone acetate will be added at a dose of 10 mg per day.
Drug: Placebo — Participants will take the placebo oral solution at a dose of 10 mL twice daily (30 minutes after breakfast and dinner). The placebo intervention will commence immediately after the cessation of menstruation and will continue until the onset of the subsequent menstrual period. At the completion of each menstrual cycle, the treatment will be resumed. Each treatment course will last for 28 days, with a total of three consecutive cycles administered.
  Arms: Placebo + Hormone replacement therapy

SUMMARY:
Study Summary

This clinical trial aims to evaluate the efficacy and safety of the traditional Chinese herbal formula Huanjingjian decoction in women with premature ovarian insufficiency (POI). The study is designed to address the following key questions:

1. Does Huanjingjian decoction improve clinical symptoms in patients with POI?
2. What adverse medical events, if any, occur during the treatment with Huanjingjian decoction? To answer these questions, researchers will compare Huanjingjian decoction plus hormone replacement therapy (HRT) with placebo plus HRT, in order to determine whether Huanjingjian decoction provides additional therapeutic benefits in the management of POI.

Participants will:

Receiving either Huanjingjian decoction plus HRT, or placebo plus HRT. Attending monthly clinic visits over a 6-month period for clinical assessments and laboratory testing.

Keeping a detailed diary to record symptoms, treatment adherence, and menstrual flow, as measured by the number of sanitary pads used.

DETAILED DESCRIPTION:
This study is a prospective, randomized, controlled clinical trial designed to evaluate the efficacy of the traditional Chinese herbal formula Huanjingjian decoction in combination with hormone replacement therapy for the treatment of premature ovarian insufficiency. The primary objective is to determine whether the addition of Huanjingjian decoction to hormone replacement therapy provides greater improvement in clinical symptoms compared with placebo combined with hormone replacement therapy. It is hypothesized that, at 12 weeks, treatment with Huanjingjian decoction in combination with hormone replacement therapy will result in superior clinical outcomes relative to placebo combined with hormone replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 39 years
* Meet the diagnostic criteria for Premature Ovarian Insufficiency (POI) according to the 2024 ESHRE Guideline on Premature Ovarian Insufficiency

Exclusion Criteria:

* Menstrual disorders attributable to congenital gonadal dysgenesis or acquired structural pathologies;
* Menstrual irregularities secondary to endocrine disorders, including polycystic ovary syndrome (PCOS), hyperprolactinemia, dysfunctional uterine bleeding (DUB), gonadal hormone deficiency, hyperthyroidism, and other related endocrine conditions;
* Oligomenorrhea or amenorrhea induced by surgical or medical interventions, such as chemotherapy, pelvic radiotherapy, ovarian cystectomy, ovarian drilling, ovarian wedge resection, salpingectomy, tubal ligation, pelvic abscess surgery, or uterine artery embolization;
* History of abnormal vaginal bleeding accompanied by clinically significant findings on endometrial biopsy, or unexplained irregular vaginal bleeding within the preceding 12 months;
* Suspected cervical malignancy or precancerous cervical lesions, suspected malignant breast tumors, or a known or suspected history of hormone-dependent tumors or malignancies;
* Previous or current history of deep vein thrombosis (DVT), pulmonary embolism, thrombotic disorders, or cerebrovascular events (stroke);
* Presence of uncontrolled and/or undiagnosed systemic diseases that could confound study results or compromise patient safety, including severe hepatic, renal, cardiac, or neurological disorders;
* Known hypersensitivity or allergy to any study-related medications;
* Pregnancy or lactation;
* Participation in other clinical trials within the last 3 months;
* Failure or refusal to provide written informed consent.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 276 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2030-07-30 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
Disease-Specific Quality of Life Assessment | From the time of enrollment through the 6-month follow-up period
  The Chinese version of the Menopause-Specific Quality-of-Life questionnaire (CMS) will be used to assess disease-specific quality of life. This validated instrument demonstrates high reliability, validity, and sensitivity, and is widely recognized as a comprehensive tool for evaluating the physical and psychological well-being of Chinese women during menopause.
  The CMS is self-administered and uses a Likert-scale format. Each item evaluates the impact of menopausal symptoms experienced in the past month. The CMS includes 29 items across four domains: vasomotor (3 items), psychosocial (7 items), physical (16 items), and sexual (3 items). Respondents first indicate whether a symptom is present; if endorsed, they rate its severity from 0 (not bothersome) to 6 (extremely bothersome). Each item is scored from 1 (not present) to 8 (extremely bothersome). Assessments will be conducted at baseline, 3 months, and 6 months.

SECONDARY OUTCOMES:
Changes in serum anti-Müllerian hormone (AMH) levels | From the time of enrollment through the 6-month follow-up period
  Assessments will be conducted at baseline, 3 months, and 6 months, with measurements taken on day 3 of the menstrual cycle.
Change in follicle-stimulating hormone (FSH) levels | From the time of enrollment through the 6-month follow-up period
  Assessments will be conducted at baseline, 3 months, and 6 months, with measurements taken on day 3 of the menstrual cycle.
Change in luteinizing hormone (LH) levels | From the time of enrollment through the 6-month follow-up period
  Assessments will be conducted at baseline, 3 months, and 6 months, with measurements taken on day 3 of the menstrual cycle.
Change in estradiol (E2) levels | From the time of enrollment through the 6-month follow-up period
  Assessments will be conducted at baseline, 3 months, and 6 months, with measurements taken on day 3 of the menstrual cycle.
Antral follicle count | From the time of enrollment through the 6-month follow-up period
  Antral follicle count (AFC) will be assessed by transvaginal ultrasound between days 2 and 5 of the menstrual cycle at baseline, 3 months, and 6 months. Menstruation may be spontaneous or induced with progestin; in cases of persistent amenorrhea, ovarian function assessment will be performed irrespective of the menstrual cycle.
Ovarian volume evaluation | From the time of enrollment through the 6-month follow-up period
  Ovarian volume evaluation will be assessed by transvaginal ultrasound between days 2 and 5 of the menstrual cycle at baseline, 3 months, and 6 months. Menstruation may be spontaneous or induced with progestin; in cases of persistent amenorrhea, ovarian function assessment will be performed irrespective of the menstrual cycle.
Menstrual recovery rate | From the time of enrollment through the 6-month follow-up period
  The menstrual recovery rate (%) will be calculated as follows: Menstrual Recovery Rate (%) = (Number of participants with menstrual recovery ÷ Total number of participants) × 100%. Assessment of this outcome will be conducted at 6 months.
Generic quality of life | From the time of enrollment through the 6-month follow-up period
  Generic quality of life will be assessed using the Short Form-36 Health Survey (SF-36) at baseline, 3 months, and 6 months to evaluate the overall impact of the intervention on health-related quality of life. The SF-36 is a validated and widely used instrument comprising eight domains: physical functioning, role limitations due to physical or emotional problems, bodily pain, general health, vitality, social functioning, and mental health. Scores range from 0 to 100, with higher scores indicating better perceived health status.

OTHER OUTCOMES:
Number of participants with adverse events as assessed by CTCAE v4.0 （Safety Outcome） | From the time of enrollment through the 6-month follow-up period
  All adverse events occurring throughout the intervention and follow-up periods will be recorded.
Morisky Medication Adherence Scale (MMAS-8) | From the time of enrollment through the 6-month follow-up period
  The Morisky Medication Adherence Scale (MMAS-8) is a widely used self-reported questionnaire designed to assess patients' medication adherence. The scale consists of 8 items, with a total score ranging from 0 to 8. Higher scores indicate better adherence. A score of 8 indicates high adherence, scores of 6-7 indicate medium adherence, and scores below 6 indicate low adherence. The assessment will be conducted at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: TE LIU, Doctor, Study Chair — Shanghai Geriatric Institute of Chinese Medicine
Locations (1):
- Jingan hospital of Traditional Chinese Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Primary outcome data under request
Supporting Information: Study Protocol, SAP
Time Frame: From publication until the third year after publication
Access Criteria: Research scope